CLINICAL TRIAL: NCT00542516
Title: Comparison Between Two Techniques of Volemic Expansion in Hip Replacement Arthroplasty: Hydroxyethyl Starch Versus Ringer's Lactate
Brief Title: Comparison Between Two Techniques of Volemic Expansion in Hip Replacement Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: adilson hamaji - supervisor anesthesia institute orthopedic USP, University São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC524/04
Record Dates: First submitted 2007-10-02; First posted 2007-10-11 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Hip Replacement Arthroplasty
Keywords: Hip Replacement Arthroplasty; Hydroxyethyl Starch; Hemodilution; Hetastarch; Colloids
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4; Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HES 130/04 (Experimental): Pre-expansion with HES
  Interventions: Drug: Hydroxyethyl Starch
- Ringer's lactate (Active Comparator): Pre-expansion with Ringer's lactate
  Interventions: Drug: Hydroxyethyl Starch; Drug: Ringer's lactate

INTERVENTIONS:
Drug: Hydroxyethyl Starch — Dosage: 30ml/kg; frequency: one time; duration: 60min
  Other Names: Voluven
Drug: Ringer's lactate — Dosage: 30ml/kg; frequency: one time; duration: 60min.After 10ml-kg-h both groups
  Arms: Ringer's lactate

SUMMARY:
Currently the most use solution to volemic reposition in hip replacement arthroplasty is the crystalloid solution. This trial intends to compare two different volemic replacements: HES and Ringer's lactate. This research has been analyzing hemodynamic parameters and the coagulation status before and after the pre-expansion with the solutions above mentioned.

DETAILED DESCRIPTION:
This trial is randomized an blind to the physician who is analyzing the results.It has been select adults; both sex; ASA I and II. These patients must be submitted to hip arthroplasty replacement. The anesthesia technique is single shot spinal anesthesia. Primary endpoint: assessment alternative; technique replacement volemic with HES 130/04. Secondary endpoint: haemostatic abnormalities; blood loss; transfusion blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients involved: adults, ASA I and II;
* Surgery: hip replacement arthroplasty.

Exclusion Criteria:

* Allergy starch;
* Anemia;
* Dysfunction renal;
* Heart insufficiency;
* Morbid obesity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
HES expansion plasmatic efficacy | 24 hours

SECONDARY OUTCOMES:
Blood transfusion | 24 hours
Haemostatic alterations | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: José Otávio C Auler Junior, PhD/Chairman, Study Chair — Hospital das Clínicas - Medicine School of the University of São Paulo
Locations (1):
- Institute of Orthopedics and Traumatology of HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Langeron O, Doelberg M, Ang ET, Bonnet F, Capdevila X, Coriat P. Voluven, a lower substituted novel hydroxyethyl starch (HES 130/0.4), causes fewer effects on coagulation in major orthopedic surgery than HES 200/0.5. Anesth Analg. 2001 Apr;92(4):855-62. doi: 10.1097/00000539-200104000-00011. PMID 11273914
- [Background] Gallandat Huet RC, Siemons AW, Baus D, van Rooyen-Butijn WT, Haagenaars JA, van Oeveren W, Bepperling F. A novel hydroxyethyl starch (Voluven) for effective perioperative plasma volume substitution in cardiac surgery. Can J Anaesth. 2000 Dec;47(12):1207-15. doi: 10.1007/BF03019870. PMID 11132743
- [Background] Haisch G, Boldt J, Krebs C, Kumle B, Suttner S, Schulz A. The influence of intravascular volume therapy with a new hydroxyethyl starch preparation (6% HES 130/0.4) on coagulation in patients undergoing major abdominal surgery. Anesth Analg. 2001 Mar;92(3):565-71. doi: 10.1097/00000539-200103000-00003. PMID 11226079 (Retraction: PMID 21451074 Anesth Analg. 2011 May;112(5):1225)
- [Background] Jungheinrich C, Scharpf R, Wargenau M, Bepperling F, Baron JF. The pharmacokinetics and tolerability of an intravenous infusion of the new hydroxyethyl starch 130/0.4 (6%, 500 mL) in mild-to-severe renal impairment. Anesth Analg. 2002 Sep;95(3):544-51, table of contents. doi: 10.1097/00000539-200209000-00007. PMID 12198032
- [Background] Boldt J, Suttner S. Plasma substitutes. Minerva Anestesiol. 2005 Dec;71(12):741-58. PMID 16288182
- [Background] Mielke LL, Entholzner EK, Kling M, Breinbauer BE, Burgkart R, Hargasser SR, Hipp RF. Preoperative acute hypervolemic hemodilution with hydroxyethylstarch: an alternative to acute normovolemic hemodilution? Anesth Analg. 1997 Jan;84(1):26-30. doi: 10.1097/00000539-199701000-00005. PMID 8988994
- [Background] Gandhi SD, Weiskopf RB, Jungheinrich C, Koorn R, Miller D, Shangraw RE, Prough DS, Baus D, Bepperling F, Warltier DC. Volume replacement therapy during major orthopedic surgery using Voluven (hydroxyethyl starch 130/0.4) or hetastarch. Anesthesiology. 2007 Jun;106(6):1120-7. doi: 10.1097/01.anes.0000265422.07864.37. PMID 17525586
- [Background] Otsuki DA, Fantoni DT, Margarido CB, Marumo CK, Intelizano T, Pasqualucci CA, Costa Auler JO Jr. Hydroxyethyl starch is superior to lactated Ringer as a replacement fluid in a pig model of acute normovolaemic haemodilution. Br J Anaesth. 2007 Jan;98(1):29-37. doi: 10.1093/bja/ael312. Epub 2006 Nov 26. PMID 17130138